CLINICAL TRIAL: NCT07094555
Title: The Effect of Two Different Interventions Applied During the Transfer of Children to the Operating Room for Circumcision on Fear, Anxiety, Comfort and Pain Levels: Randomized Controlled Trial
Brief Title: The Effect of Two Different Interventions Applied During the Transfer of Children to the Operating Room for Circumcision on Fear, Anxiety, Comfort and Pain Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MELİS CAN KESGİN GÜNGÖR (Other)
Responsible Party: Sponsor-Investigator, MELİS CAN KESGİN GÜNGÖR, Principal Investigator, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 81822950.903/142
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Male Circumcision
Keywords: Pain; Anxiety; Child; Kaleidoscope; Comfort; Fear; Animal Assisted Practice
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal Assisted Practice Group (Experimental)
  Interventions: Behavioral: Animal Assisted Practice
- Kaleidoscope Group (Experimental)
  Interventions: Behavioral: Kaleidoscope
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Animal Assisted Practice — The animal-assisted intervention group initiated interaction with a goldfish in a portable aquarium during the preoperative period and accompanied them until they reached the operating room.
  Arms: Animal Assisted Practice Group
Behavioral: Kaleidoscope — The kaleidoscope group was distracted with a kaleidoscope during the preoperative period and continued this intervention until they reached the operating room.
  Arms: Kaleidoscope Group

SUMMARY:
The aim of this randomized controlled experimental study was to determine the effects of two different interventions on fear, anxiety, comfort, and pain levels during the transfer of children undergoing circumcision to the operating room.

The main questions it aims to answer are:

* H1: Animal-assisted intervention during transfer to the operating room affects children's fear.
* H2: Animal-assisted intervention during transfer to the operating room affects children's anxiety.
* H3: Animal-assisted intervention during transfer to the operating room affects children's comfort.
* H4: Animal-assisted intervention during transfer to the operating room affects children's pain.
* H5: Playing with a kaleidoscope during transfer to the operating room affects children's fear.
* H6: Playing with a kaleidoscope during transfer to the operating room affects children's anxiety.
* H7: Playing with a kaleidoscope during transfer to the operating room affects children's comfort.
* H8: Playing with a kaleidoscope during transfer to the operating room affects children's pain.

Researchers will investigate the effects of animal-assisted intervention and kaleidoscopes on anxiety, fear, pain, and comfort during the transfer to the operating room in boys aged 7-10 undergoing circumcision. A comparison will be made with a control group to determine this effectiveness.

Participants:

* The animal-assisted intervention group will initiate interaction with a goldfish in a portable aquarium during the preoperative period and accompany them until they arrive in the operating room.
* The kaleidoscope group will be distracted with a kaleidoscope during the preoperative period and continue this intervention until they arrive in the operating room.
* The control group will follow the hospital's routine patient transfer procedure.

ELIGIBILITY:
Inclusion Criteria:

* 7-10 age group
* Circumcision performed under general anesthesia or sedation
* Pain level 0 before surgery
* Child has literacy skills
* Child and parent volunteer to participate in the study

Exclusion Criteria:

* The child has had previous surgical experience
* The child is allergic to fish products or fish meal
* The child has a special condition that may cause difficulty understanding and perceiving
* Any complications develop in the postoperative period
* The child and parent wish to withdraw from the study
* The child's hemodynamic instability

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — male
Enrollment: 90 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Animal-assisted therapy intervention applied during transfer to the operating room changes Child Anxiety Scale scores in the preoperative period. | 10 minutes before surgery
  Child Anxiety Scale: The score that can be obtained from the scale varies between 0 and 10 points. As the score increases, the anxiety level also increases.
Animal-assisted therapy intervention applied during transfer to the operating room changes Child Fear Scale scores in the preoperative period. | 10 minutes before surgery
  Child Fear Scale: The score that can be obtained from the scale varies between 0 and 4 points. As the score increases, the fear level also increases.
Animal-assisted therapy intervention applied during transfer to the operating room changes Wong-Baker pain scale scores in the postoperative period. | up to the 1st postoperative hour
  Wong-Baker Pain Scale: The score that can be obtained from the scale varies between 0 and 10 points. As the score increases, the pain level also increases.
Animal-assisted therapy intervention applied during transfer to the operating room changes Comfort Behaviors Checklist scores in the postoperative period. | up to the 1st postoperative hour
  Comfort Behaviors Checklist: The score that can be obtained from the scale varies between 25 and 100 points. As the score increases, the comfort level also increases.
Kaleidoscope intervention applied during transfer to the operating room changes Child Anxiety Scale scores in the preoperative period. | 10 minutes before surgery
  Child Anxiety Scale: The score that can be obtained from the scale varies between 0 and 10 points. As the score increases, the anxiety level also increases.
Kaleidoscope intervention applied during transfer to the operating room changes Child Fear Scale scores in the preoperative period. | 10 minutes before surgery
  Child Fear Scale: The score that can be obtained from the scale varies between 0 and 4 points. As the score increases, the fear level also increases.
Kaleidoscope intervention applied during transfer to the operating room changes Wong-Baker pain scale scores in the postoperative period. | up to the 1st postoperative hour
  Wong-Baker Pain Scale: The score that can be obtained from the scale varies between 0 and 10 points. As the score increases, the pain level also increases.
Kaleidoscope intervention applied during transfer to the operating room changes Comfort Behaviors Checklist scores in the postoperative period. | up to the 1st postoperative hour
  Comfort Behaviors Checklist: The score that can be obtained from the scale varies between 25 and 100 points. As the score increases, the comfort level also increases.

IPD SHARING:
Plan to Share IPD: No